CLINICAL TRIAL: NCT04329390
Title: MAC Project, Monitoring of AntiCoagulant Therapies (MAC)
Acronym: MAC
Status: Completed | Type: Observational
Sponsor: Quovadis Associazione (Other)
Responsible Party: Sponsor
Other Study IDs: MAC Project
Record Dates: First submitted 2020-03-09; First posted 2020-04-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Anticoagulants and Bleeding Disorders
Keywords: anticoagulant; DOAC; OAC; benefit-risk
MeSH Terms: conditions — Hemostatic Disorders | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anticoagulant: Subjects of both sexes, aged 18 years or older, requiring the prescription of, or already on oral anticoagulant treatment, will be eligible for the study, irrespective of the index event, of the intended treatment duration, and the type of drug used.
  Interventions: Drug: Anticoagulant drugs

INTERVENTIONS:
Drug: Anticoagulant drugs — Prescription of, or already on oral anticoagulant treatment.
  Other Names: OAC

SUMMARY:
MAC Project is a prospective cohort, multicenter, observational, no-profit study aimed to prospectively collect reliable real-life clinical information in unselected VTE or NVAF patients treated with any DOAC, during a medium-long term follow-up period.

DETAILED DESCRIPTION:
MAC Project is a prospective cohort, multicenter, observational, no-profit study aimed to prospectively collect reliable real-life clinical information in unselected VTE or NVAF patients treated with any DOAC, during a medium-long term follow-up period. Patients will be investigated in Italian hospital-based clinical centers, skilled in the management of adult patients with VTE or NVAF requiring anticoagulant treatment, and followed-up up to 5 years. The drugs will be prescribed according to current standards of care and regulations and not provided by any sponsor. The primary outcome is to collect and evaluate the safety and efficacy data of DOACs in a real-life setting, regardless of the underlying pathology, and the duration of treatment. The secondary outcome is to separately evaluate safety and efficacy of DOACs for treatment of cardiovascular diseases, specifically considering treatment duration, as follows: short-term (e.g., superficial venous thrombosis); medium-term (e.g., deep vein thrombosis, pulmonary embolism, etc.); long-term (e.g., atrial fibrillation, prevention of recurrent VTE or long-term treatment of recurrent VTE, peripheral arterial obstructive disease, etc.).Investigators will store event-driven clinical information into a REDCap based on-line EDC system about management and outcome of all efficacy and safety end-points; treatment compliance/adherence; VTE risk factors; thromboembolic and haemorrhagic risk-scores; comorbidities; concomitant treatments; patients' appreciation by a specific score (ACTS); clinical or adverse events; survival; possible causes of death.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years,
* mandatory anticoagulant treatment
* ability to understand the purposes of the study
* ability to express valid informed consent.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting: clinical centers, either hospital-based or outpatient clinics, experienced in the management of patients with cardiovascular diseases requiring anticoagulant treatment, either on short- (e.g., superficial venous thrombosis), medium- (e.g., deep-vein thrombosis, pulmonary embolism, acute coronary syndrome, etc.), and long-term (e.g., atrial fibrillation, mechanic heart valves, secondary prevention of recurrent VTE, obstructive arterial disease of the lower limbs, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
SAFETY OF OAC THERAPY | 5 years
  incidence of major bleeding, incidence of clinically relevant non-major bleeding, incidence of minor bleeding, incidence of serious adverse events, incidence of mortality (VTE-related, cardiovascular, and all-cause).
EFFICACY OF OAC THERAPY | 5 years
  incidence of symptomatic recurrent VTE, incidence of symptomatic recurrent VTE in the various treatment subgroups, incidence of stroke (ischemic and haemorrhagic), incidence of systemic embolic events, number of hospital admissions related to cardiovascular (either venous or arterial) disease, incidence of post-thrombotic syndrome.

SECONDARY OUTCOMES:
Time relate outcomes | 5 years
  To separately evaluate safety and efficacy of DOACs for treatment of cardiovascular diseases, specifically considering treatment duration, as follows: short-term (e.g., superficial venous thrombosis); medium-term (e.g., deep vein thrombosis, pulmonary embolism, etc.); long-term (e.g., atrial fibrillation, prevention of recurrent VTE or long-term treatment of recurrent VTE, peripheral arterial obstructive disease, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Bortoluzzi, MD, Principal Investigator — Quovadis Associazione
Locations (1):
- Giuseppe Camporese, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04329390/Prot_000.pdf